CLINICAL TRIAL: NCT04790279
Title: Amlodipine Versus Nifedipine ER for the Management of Postpartum Hypertension: A Randomized Controlled Noninferiority Trial
Brief Title: Amlodipine Versus Nifedipine ER for the Management of Postpartum Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00106643
Record Dates: First submitted 2021-03-03; First posted 2021-03-10 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2022-12

CONDITIONS: Hypertension in Pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Amlodipine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Amlodipine (Experimental)
  Interventions: Drug: Amlodipine
- Nifedipine ER (Active Comparator)
  Interventions: Drug: NIFEdipine ER

INTERVENTIONS:
Drug: Amlodipine — Initiation of amlodipine 2.5 mg
  Arms: Amlodipine
Drug: NIFEdipine ER — Initiation of nifedipine ER 30 mg
  Arms: Nifedipine ER

SUMMARY:
A significant number of pregnancies are complicated by hypertensive disorders. Hypertension often worsens in the postpartum period and many women need started on medications. Currently, recommended medications for blood pressure management in pregnant and postpartum women are limited, with labetalol and nifedipine ER being the most commonly used medications. While these medications are both effective, they are not without limitations. Amlodipine is a medication in the same class as nifedipine ER. It is a first-line antihypertensive in the general population. It tends to have less side effects than nifedipine ER. It has not been studied specifically in postpartum women. The purpose of this study is to determine if amlodipine is noninferior to nifedipine ER in managing hypertension in the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women with a diagnosis of chronic hypertension, gestational hypertension, or preeclampsia
* Delivery at or beyond 20 weeks' gestation
* Need for antihypertensive therapy, defined as blood pressure >/= 150 mmHg systolic and/or 100 mmHg diastolic on two occasions four hours apart or isolated blood pressure >160/110 mmHg
* English or Spanish-speaking
* Age 18 years or older

Exclusion Criteria:

* Use of antihypertensive prior to delivery (for any indication)
* Allergy to nifedipine ER or amlodipine
* Persistent tachycardia (as defined by the treatment team)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katelyn Pratt, MD, Study Chair — Prisma Health
Locations (1):
- Greenville Memorial Hospital, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Background] ACOG Practice Bulletin No. 202: Gestational Hypertension and Preeclampsia. Obstet Gynecol. 2019 Jan;133(1):1. doi: 10.1097/AOG.0000000000003018. PMID 30575675
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 203: Chronic Hypertension in Pregnancy. Obstet Gynecol. 2019 Jan;133(1):e26-e50. doi: 10.1097/AOG.0000000000003020. PMID 30575676
- [Background] Ainuddin J, Javed F, Kazi S. Oral labetalol versus oral nifedipine for the management of postpartum hypertension a randomized control trial. Pak J Med Sci. 2019 Sep-Oct;35(5):1428-1433. doi: 10.12669/pjms.35.5.812. PMID 31489020
- [Background] Magee L, von Dadelszen P. Prevention and treatment of postpartum hypertension. Cochrane Database Syst Rev. 2013 Apr 30;2013(4):CD004351. doi: 10.1002/14651858.CD004351.pub3. PMID 23633317
- [Background] Cairns AE, Pealing L, Duffy JMN, Roberts N, Tucker KL, Leeson P, MacKillop LH, McManus RJ. Postpartum management of hypertensive disorders of pregnancy: a systematic review. BMJ Open. 2017 Nov 28;7(11):e018696. doi: 10.1136/bmjopen-2017-018696. PMID 29187414
- [Background] Sharma KJ, Greene N, Kilpatrick SJ. Oral labetalol compared to oral nifedipine for postpartum hypertension: A randomized controlled trial. Hypertens Pregnancy. 2017 Feb;36(1):44-47. doi: 10.1080/10641955.2016.1231317. Epub 2016 Oct 27. PMID 27786578
- [Background] 8. Bloch, M. (2020). In Basile J. (Ed.), Major side effects and safety of calcium channel blockers. UpToDate.
- [Background] Hosie J, Bremner AD, Fell PJ, James IG, Saul PA, Taylor SH. Comparison of early side effects with amlodipine and nifedipine retard in hypertension. Cardiology. 1992;80 Suppl 1:54-9. doi: 10.1159/000175048. PMID 1534716
- [Background] Naito T, Kubono N, Deguchi S, Sugihara M, Itoh H, Kanayama N, Kawakami J. Amlodipine passage into breast milk in lactating women with pregnancy-induced hypertension and its estimation of infant risk for breastfeeding. J Hum Lact. 2015 May;31(2):301-6. doi: 10.1177/0890334414560195. Epub 2014 Dec 1. PMID 25447596

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were randomized at the time of enrollment. Only patients meeting pre-defined criteria were started on an anti-hypertensive.
Period: Overall Study
Arm/Group | Amlodipine | Nifedipine ER
Started | 87 | 88
Completed | 51 | 69
Not Completed | 36 | 19
Not completed — Did not meet medication start criteria | 27 | 15
Not completed — Required long acting antihypertensive intrapartum | 1 | 0
Not completed — Protocol Violation | 8 | 3
Not completed — Developed complication requiring alternative regimen | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Amlodipine: Patients randomized to amlodipine
- Nifedipine ER: Patients randomized to nifedipine ER
- Total: Total of all reporting groups
Arm/Group | Amlodipine | Nifedipine ER | Total
Number analyzed (Participants) | 87 | 88 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (6.8) | 27.8 (5.9) | 27.8 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data were not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 87 | 88 | 175
BMI at delivery [Mean (Standard Deviation); unit: kg/m2] | 36.8 (9.3) | 37.0 (10.1) | 36.9 (9.7)
Parity [Median (Full Range); unit: number of deliveries] | 1 [0 to 9] | 1 [0 to 5] | 1 [0 to 9]
Gestational age at delivery [Mean (Standard Deviation); unit: weeks] | 35.7 (2.5) | 35.6 (3.3) | 35.6 (2.9)
Mode of delivery [Number; unit: participants]
  Vaginal | 40 | 44 | 84
  Cesarean | 47 | 44 | 91
Hypertensive diagnosis [Number; unit: participants] — May have more than 1 diagnosis
  participants
    Chronic hypertension | 21 | 22 | 43
    Preeclampsia without severe features | 3 | 3 | 6
    Preeclampsia with severe features | 84 | 81 | 165
Diabetes [Count of Participants; unit: Participants]
  None | 71 | 66 | 137
  Gestational | 8 | 15 | 23
  Pre-gestational | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay
Description: length of stay from delivery until discharge
Time Frame: Through hospital stay, on average 2-5 days
Population: Amlodipine Intent To Treat
Measure: Median (95% Confidence Interval); unit: hours
Groups:
- Amlodipine: Amlodipine Intent to Treat
- Nifedipine ER: Nifedipine ER Intent To Treat
Arm/Group | Amlodipine | Nifedipine ER
Number analyzed (Participants) | 87 | 88
hours | 73.5 [67.0 to 81.0] | 72.0 [66.5 to 78.5]

2. Secondary Outcome: Number of Acute Treatments After Medication Initiation
Time Frame: Through hospital stay, on average 2-5 days
Population: Patients who received at least 1 dose of assigned study medication at correct starting dose
Measure: Median (Standard Deviation); unit: number acute treatments
Groups:
- Amlodipine: Amlodipine Per Protocol
- Nifedipine ER: Nifedipine ER Per Protocol
Arm/Group | Amlodipine | Nifedipine ER
Number analyzed (Participants) | 51 | 69
number acute treatments | 4.0 (2.7) | 1.5 (1.5)

3. Secondary Outcome: Patient Reported Side Effects
Description: Side effects based on patient reported survey where 1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5 = always
Time Frame: Through hospital stay, on average 2-5 days
Population: Patients receiving at least 1 dose of assigned study medication at correct starting dose
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Amlodipine | Nifedipine ER
Number analyzed (Participants) | 51 | 69
score on a scale
  Flushing | 1.33 (0.72) | 1.60 (1.00)
  Swelling | 1.55 (1.16) | 1.71 (1.09)
  Headaches | 1.71 (1.06) | 1.98 (1.17)
  Other | 1.24 (0.85) | 1.11 (0.55)

4. Secondary Outcome: Number of Patients Discontinuing Medication Due to Side Effects
Time Frame: Through hospital stay, on average 2-5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Amlodipine | Nifedipine ER
Number analyzed (Participants) | 51 | 69
Participants | 0 | 7

5. Secondary Outcome: Number of Patients Requiring Hospital Readmission
Time Frame: until 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Amlodipine | Nifedipine ER
Number analyzed (Participants) | 51 | 69
Participants | 3 | 3

6. Secondary Outcome: Breastfeeding Duration of 6+ Weeks
Time Frame: until 6 weeks postpartum
Population: Only includes patients who answered relevant question on breastfeeding questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Amlodipine | Nifedipine ER
Number analyzed (Participants) | 12 | 17
Participants | 4 | 3

7. Secondary Outcome: Number of Patients Reporting Satisfaction With Breastfeeding Experience on Patient-completed Questionnaire
Time Frame: until 6 weeks postpartum
Population: Only includes patients who answered relevant question on breastfeeding questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Amlodipine | Nifedipine ER
Number analyzed (Participants) | 27 | 36
Participants | 22 | 32

ADVERSE EVENTS:
Time Frame: Through 6 weeks postpartum
Description: Only patients receiving at least one dose of assigned study medication are included
Arm/Group | Amlodipine | Nifedipine ER
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/69
Serious Adverse Events (participants affected / at risk) | 4/53 | 4/69
Other Adverse Events (participants affected / at risk) | 19/53 | 26/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amlodipine (N=53) | Nifedipine ER (N=69)
Readmission (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3)
Prolonged hospitalization (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amlodipine (N=53) | Nifedipine ER (N=69)
Prolonged hospitalization (Pregnancy, puerperium and perinatal conditions) | 14 | 11
Side effect requiring discontinuation (Pregnancy, puerperium and perinatal conditions) | 0 | 7
Triage/ER visit (Pregnancy, puerperium and perinatal conditions) | 5 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT04790279/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT04790279/ICF_001.pdf